CLINICAL TRIAL: NCT03087812
Title: Durability of Flexible Ureteroscopes and Causes of Infection During Flexible Ureterorenoscopy
Status: Completed | Type: Observational
Sponsor: Clinical Research Office of the Endourological Society (Other)
Responsible Party: Sponsor
Other Study IDs: NL201501
Record Dates: First submitted 2015-11-19; First posted 2017-03-23 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Kidney Stones
Keywords: Microbiological burden; kidney; stone; durability of flexible endoscopes
MeSH Terms: conditions — Kidney Calculi; Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study in which data on consecutive patients who undergo ureterorenoscopy with the use of a flexible ureterorenoscope are collected. In total 20 new ureteroscopes are usedfrom Olympus andfrom Storz) to study the durability of the ureteroscopes and the possible microbiological load.

DETAILED DESCRIPTION:
This is an observational study in which data on consecutive patients who undergo ureterorenoscopy with the use of a flexible ureterorenoscope are collected. In total 6 new ureteroscopes are used (3 from Olympus and 3 from Storz) to study the durability of the ureteroscopes and the possible microbiological load.

Before the procedure is started the endoscope is tested for its microbiological load in two different ways:1. Shake the tip of the flexible ureterorenoscope 5 seconds in a sterile container filled with 10 cc of NaCl 0.9% 2. Flush the working channel of the ureterorenoscope with 10 cc of NaCl 0.9% and collect the sample in a sterile container.

After the procedure is finished, the endoscope is tested for its microbiological load in two different ways:

1. Shake the tip of the flexible ureterorenoscope 5 seconds in a sterile container filled with 10 cc of NaCl 0.9% 2. Flush the working channel of the ureterorenoscope with 10 cc of NaCl 0.9% and collect the sample in a sterile container.

Transfer all samples to the lab as soon as possible but at least within four hours after collecting the samples.

As for the clinical efficacy during each procedure a detailed questionnaire about the use of each ureteroscope is filled out. This includes the ease of use making mention on quality of the image, torque, flexibility and durability.

Data will be collected through electronic case report forms (eCFRs), with use of an online Data Management system (DMS).

ELIGIBILITY:
Inclusion Criteria:

* Patient presented with a diagnosis to undergo a ureterorenoscopy using a flexible ureterorenoscope
* over 18 years
* has signed informed consent
* the patient is being treated with the designated flexible ureterorenoscope

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population compromises those patients of over eighteen years old diagnosed to undergo a ureterorenoscopy (diagnostic or therapeutic) with a flexible ureterorenoscope.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Microbiological load | 2 years
  To evaluate the pre-operative microbiological load of the tip and the working channel of the most common used flexible ureteroscopes, after high level disinfection

SECONDARY OUTCOMES:
Durability | 2 years
  To evaluate the durability of the most common used flexible ureteroscopes in terms of number of procedures, total use time and total degrees of flexibility loss until the first repair is needed.
Factors affecting durability | 2 years
  To evaluate descriptive data on factors that may affect the durability of the flexible ureteroscopes. Factors measured are treatment time, treatment indication and anatomical location in the urinary tract, method of ureteroscope insertion number and type of accessory instrumentation through the working channel, difference in users, number of forcing the scope during the procedure and the number of disinfections.

CONTACTS AND LOCATIONS:
Overall Officials: Jean de la Rosette, MD, PhD, Study Chair — Clinical Research Office of the Endourological Society
Locations (1):
- AMC University Hospital, Amsterdam, Netherlands